CLINICAL TRIAL: NCT04077957
Title: Treat-to-target Strategy in Ankylosing Spondylitis Using Etanercept and Conventional Synthetic DMARDs, a Prospective Randomized Controlled Study
Brief Title: Treat-to-target Strategy in Ankylosing Spondylitis Using Etanercept and Conventional Synthetic DMARDs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2019-122
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Ankylosing Spondylitis; Spondyloarthritis
Keywords: disease modifying anti-rheumatic drugs(DMARDs); etanercept; ankylosing spondylitis; spondyloarthritis; treat-to-target
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis | interventions — Methotrexate; Sulfasalazine; Hydroxychloroquine; Etanercept; Anbainuo protein, human

STUDY DESIGN:
Intervention Model Description: All enrolled participants will be randomly divided into 2 groups evenly. Participants in Group 1 will be treated with etanercept and conventional synthetic DMARDs based on treat-to-target strategy, while the others in Group 2 will be treated with conventional therapy scheme using etanercept only.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1. Experimental (Experimental): Etanercept 50mg per week plus conventional synthetic DMARDs(csDMARDs, methotrexate 10mg per week, sulfasalazine 2.25g per day, hydroxychloroquine 0.2g per day) for 4 weeks when in high disease activity; etanercept 50mg per week plus csDMARDs for 2 weeks and continue with csDMARDs only for 2 weeks when in low disease activity; csDMARDs only for 4 weeks when in disease remission status.
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Hydroxychloroquine; Drug: Etanercept (50mg per week, for 4 weeks); Drug: Etanercept (50mg per week, for 2 weeks)
- Group 2. Positive Control (Active Comparator): Etanercept 50mg per week for first 12 weeks; etanercept 50mg per ten days for second 12 weeks; etanercept 25mg per week for next 12 weeks; etanercept 25mg per two week for next 12 weeks.
  Interventions: Drug: Etanercept (50mg per week)

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 10mg per week will be the background therapy in participants in Group 1. Experimental.
  Arms: Group 1. Experimental
Drug: Sulfasalazine — Sulfasalazine 2.25g per day will be the background therapy in participants in Group 1. Experimental.
  Arms: Group 1. Experimental
Drug: Hydroxychloroquine — Hydroxychloroquine 0.2g per day will be the background therapy in participants in Group 1. Experimental.
  Arms: Group 1. Experimental
Drug: Etanercept (50mg per week, for 4 weeks) — Participants in Group 1. Experimental who satisfied the criteria for high disease activity (ASDAS≥2.1) at every follow-up point will receive etanercept (50mg per week, for 4 weeks) in the next 4 weeks.
  Other Names: Anbainuo®
  Arms: Group 1. Experimental
Drug: Etanercept (50mg per week, for 2 weeks) — Participants in Group 1. Experimental who satisfied the criteria for low disease activity (2.1>ASDAS≥1.3) at every follow-up point will receive etanercept (50mg per week, for 4 weeks) in the next 2 weeks.
  Other Names: Anbainuo®
  Arms: Group 1. Experimental
Drug: Etanercept (50mg per week) — Participants in Group 2. Positive Control will receive etanercept (50mg per week, for 12 weeks) for 48 weeks.
  Other Names: Anbainuo®
  Arms: Group 2. Positive Control

SUMMARY:
This study evaluates clinical responses and cost-effectiveness of using etanercept (ETN) and conventional synthetic Disease modifying anti-rheumatic drugs (csDMARDs) with treat-to-target strategy in ankylosing spondylitis patients. Half of participants will be used treat-to-target strategy with ETN and csDMARDs, while the others will be used conventional therapy scheme with ETN only.

DETAILED DESCRIPTION:
The tumor necrosis factor inhibitors(TNFi) like etanercept(ETN) has been always recommended as the primary treatment option for active AS. But when sustained applied in daily clinical practices, it is unaffordable for patients in developing countries in most cases due to the high expense of TNFi. On this ground, this study proposes a new scheme dividing AS treatment into relatively active phase and relatively stable phase, and sequentially introducing TNFi and conventional synthetic Disease modifying anti-rheumatic drugs (csDMARDs) in each phase respectively. Taking full advantages of the rapid and precise efficacy of TNFi when short-term application in active AS and then csDMARDs combination was prescribed to maintain the remission cause by TNFi. Drug regimes are adjusted according to the different responses of individual patient based on treat-to-target strategy. TNFi is reintroduced if there is a reactive tendency and then switching to csDMARDs again when patients are in remission. Thus, the continuous low activity or remission of AS may be promising through this treating management and the treatment cost will reduce for csDMARDs partially replace TNFi in the management of relatively stable phase.

This study is designed as a prospective randomized, positive controlled, 48-week clinical trial, involving 100 patients with active ankylosing spondylitis. All enrolled patients will randomly assign to 2 groups for the comparison of the clinical responses and cost-effectiveness of our treatment scheme with that of the conventional therapy scheme of TNFi (etanercept). Multiple clinical indexes will be measured to evaluate the therapeutic effect, including Patient's Global Assessment, BASDAI and ASDAS-CRP for disease activity, BASFI for functional state, EQ-5D and SF-36 for quality-of-life assessment, SPARCC and SPARCC Sacroiliac Joint Structural Score (SSS) for sacroiliac joint invasion. We expect to assess the feasibility of our new treatment scheme in AS disease controlling and cost-effectiveness improving through this one-year follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Capability to understand and voluntarily give written informed consent that is signed and dated, before any specific procedure of the protocol is performed.
* Patients 18 to 45 years of age.
* Proven AS according to the modified New York criteria.
* Acute phase of disease with ASDAS score ≥1.3.
* Ability to reconstitute the drug and self-inject it or have a person who can do so.
* Ability to store injectable test article at 2º to 8º C.

Exclusion Criteria:

* Patients with a history of active tuberculosis, hepatitis, gastrointestinal hemorrhage, tumors, infectious diseases or combined with other rheumaimmune systemic diseases or osteoarthritis diseases.
* Pregnancy/lactation.
* Receipt of any live (attenuated) vaccines within 4 weeks before the screening visit.
* Significant concurrent medical diseases including uncompensated congestive heart failure (NYHA III-IV), myocardial infarction within 12 months, stable or unstable angina pectoris, uncontrolled hypertension, severe pulmonary disease, history of human immunodeficiency virus (HIV) infection.
* Participation in trials of other investigational medications within 30 days of entering the study.
* Clinical examination showing significant abnormalities of clinical relevance.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-07 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-07-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Assessment in Ankylosing Spondylitis 20 (ASAS-20) Response | Week 12, 24, 36, 48
  ASAS measures symptomatic improvement in AS participants. ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 20= at least >= 20 percent improvement from baseline and an absolute change >=1 unit on a 0-10 numeric scale (0=no disease activity; 10=high disease activity) in at least 3 of the domains (on a 0-10 numerical scale): Global assessment of disease activity by participant, participant's global pain intensity, function measured by BASFI and inflammation measured by the average of the last two Likert-scales in BASDAI concerning morning stiffness intensity and duration and no worsening in the remaining domain.
Percentage of Participants With Assessment in Ankylosing Spondylitis 40 (ASAS-40) Response | Week 12, 24, 36, 48
  ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants. ASAS =4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 40= at least (>=) 40 percent improvement from baseline and an absolute change >=2 unit on a 0-10 numeric scale (0=no disease activity; 10=high disease activity) in at least 3 of the domains (on a 0-10 numerical scale): Global assessment of disease activity by participant, participant's global pain intensity, function measured by BASFI and inflammation measured by the average of the last two Likert-scales in BASDAI concerning morning stiffness intensity and duration and no worsening in the remaining domain.

SECONDARY OUTCOMES:
Mean Change From Baseline in C-Reactive Protein (CRP) | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
  The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Mean Change From Baseline in Erythrocyte Sedimentation Rate (ESR) | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
  ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter/hour (mm/hr). A higher rate is consistent with inflammation.
Mean Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score | Baseline, Week 12, 24, 36, 48
  The BASDAI score was determined using a simple, self-reported questionnaire that consists of 6 questions on disease activity. Each question is scored from 0 to 10 (0 = no symptoms, 10 = very severe symptoms).
Mean Change From Baseline in Ankylosing Spondylitis Disease Activity (ASDAS) Score | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
  The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation. The questionnaire covers disease activity, back pain, and peripheral pain/swelling assessed on a visual analogue scale (from 0 (normal) to 10 (extreme pain or disability) cm) and duration of morning stiffness on a numerical rating scale (from 0 to 10, with 0 being none and 10 representing a duration of 2 hours or longer). The laboratory parameter is a measurement of C-reactive protein (mg/L) (CRP) or erythrocyte sedimentation rate (mm/h) (ESR). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and either CRP or ESR values) are combined to yield a score ranging from 0 to no defined upper limit. Higher scores indicate higher disease activity. Remission is defined as ASDAS score <1.3. Clinically important improvement is defined as a change >= 1.1 units, and major improvement is defined as a change >= 2.0 units.
Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Score | Baseline, Week 12, 24, 36, 48
  BASFI is a validated self assessment tool that determines the degree of functional limitation in AS. Participants answered 10 questions, consisting of 8 specific questions regarding function in AS and 2 questions reflecting the participant's ability to cope with everyday life. Each question was answered on a 0-10 scale (0 being no problem and 10 being the worst problem), the sum of which (divided by 10) resulted in the BASFI score (0-10).
Mean Change From Baseline in Euro Quality of Life-5 Dimensions (EQ-5D) Score | Baseline, Week 12, 24, 36, 48
  EQ 5D is a participant rated questionnaire to assess health-related quality of life. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (extreme problems).
Mean Change From Baseline in Short Form-36 Health Survey (SF-36) Score | Baseline, Week 12, 24, 36, 48
  The Medical Outcome Study health measure SF-36 questionnaire is a well-validated and widely used quality-of-life instrument. It is a self-administered survey that consists of 8 multi-item scales: The 4 subscales of the SF-36 comprises the PCS (physical functioning, role-physical, bodily pain, and general health) score and the 4 subscales of the SF-36 comprises the MCS (vitality, social functioning, role-emotional, and mental health) score. PCS and MCS are scored from 0 to 100 with higher scores indicating better health (worst value is 0 and best value is 100), which are scored using a norm-based system where linear transformations are performed to transform scores to a mean of 50 and standard deviation of 10.
Mean Change From Baseline in SpondyloArthritis Research Consortium of Canada (SPARCC) Score for the Sacroiliac Joint | Baseline, Week 4, 12, 24, 48
  SPARCC score for the sacroiliac joint was based on 6 consecutive coronal slices from posterior to anterior. Each joint was divided into 4 quadrants. Each quadrant was assigned a score of 0 = no lesion/1 = increased signal. For each slice, the score is increased by 1 for each joint that exhibits an intense signal in any quadrant. Also, for each slice, an additional score of 1 will be given for each joint that includes a lesion demonstrating continuous increased signal of a depth ≥1 cm from the articular surface. The maximum possible score is 72.
Percentage of Participants with Serious Adverse Events (SAEs) or Adverse Events (AEs) by Co-morbidity From Baseline | Baseline, Week 12, 24, 36, 48
  Any untoward medical occurrence in a participant who received study regents was considered an AE, without regard to possibility of relationship. An AE resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a SAE: death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Xiao, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No